CLINICAL TRIAL: NCT01188837
Title: The Relative Effectiveness of Three Full Kinetic Chain Treatment Protocols for Osteoarthritis of the Knee: Manual Therapy, Rehabilitation and a Combination Thereof
Brief Title: Comparing Manipulation, Rehabilitation and Combination of the Two in the Treatment of Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cleveland Chiropractic College (Other)
Collaborators: Durban University of Technology (Other); Murdoch University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-CCC08132010
Record Dates: First submitted 2010-08-24; First posted 2010-08-26 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-08

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis, Knee; Manipulation Therapy
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Full Kinetic Chain Manipulative Therapy (Active Comparator)
  Interventions: Other: Full Kinetic Chain Manipulative Therapy
- Full Kinetic Chain Rehabilitation (Active Comparator)
  Interventions: Other: Full Kinetic Chain Rehabilitation
- Full Kinetic Chain Manipulative Therapy with Rehabilitation (Active Comparator)
  Interventions: Other: Full Kinetic Chain Manipulative Therapy with Rehabilitation

INTERVENTIONS:
Other: Full Kinetic Chain Manipulative Therapy — Treatment will focus on restoring knee flexion and extension by lesser grades of mobilization and patellar mobilization along with careful high velocity low amplitude axial elongation of the knee joint.
  Additionally, manipulative therapy will be applied where needed to the full kinetic chain using diversified techniques, such as HVLA manipulation or mobilization.
  This group will receive a total of 6 treatments over a 3 week period. Outcome measures will be taken at baseline, prior to the 4th treatment and at the one week follow-up. A 3 month follow-up will be done by mail, phone or email.
  Arms: Full Kinetic Chain Manipulative Therapy
Other: Full Kinetic Chain Rehabilitation — Rehabilitative therapy includes exercises, focused soft tissue treatment and stretch to the knee and the full kinetic chain where needed based upon functional assessment. Also included; patient advice, education and home exercise recommendations for managing their KOA.
  This group will receive a total of 6 treatments over a 3 week period. Outcome measures will be taken at baseline, prior to the 4th treatment and at the one week follow-up. A 3 month follow-up will be done by mail, phone or email.
  The rehabilitative therapy group will be required to attend the initial treatment/training, the 4th visit and 1 week follow-up. Treatments 2, 3, 5 and 6 are considered optional; they may be done at home
  Arms: Full Kinetic Chain Rehabilitation
Other: Full Kinetic Chain Manipulative Therapy with Rehabilitation — This arm is a combination of the manipulative therapy arm and the rehabilitative therapy arm.
  This group receives 6 treatments over a 3 week period with a one week follow-up on site and a 3 month follow-up by mail, phone or email.
  Arms: Full Kinetic Chain Manipulative Therapy with Rehabilitation

SUMMARY:
Common medical therapies for knee osteoarthritis are patient education, drug and physical therapy, exercise and surgery. These modalities may offer improvement but drugs and surgery carry significant risk. Manipulative therapy for KOA gives pain relief and increased function. However, research suggests addition of manipulative and soft tissue therapy (to the entire kinetic chain: lumbosacral, sacroiliac, hip, knee, ankle and foot joints), may give a better outcome. Exercise therapy is considered an effective and standard care for KOA.

DETAILED DESCRIPTION:
Patients seek treatment from chiropractors for osteoarthritis (OA) and Knee OA (KOA). Significant KOA impacts 10 % of individuals aged ≥63 particularly with radiographic changes; and by age 65, 80% have these x-ray changes. KOA may be the largest cause of decreased mobility, function, disability and pain in people aged ≥ 50 in the US. KOA causes 30% > age 60 to experience decreased social activities of daily living, increased cardiovascular risk, increased fall risk and secondary depression. Overall KOA prevalence is 4% in young adults, 85% in those > 75. Beyond great personal suffering - in the US, annual financial costs associated with OA were $60 billion per year in 2000 and, for all OA and rheumatic disease $128 billion in 2003. Estimates in 2005 were 27 million people suffer significantly due to OA and by 2020 in the US and other developed nations > 12 million will suffer serious, and 19 million minor to moderate work or activity related disability from OA and KOA, with the highest prevalence expected in women.

Medical care commonly prescribed for KOA is lifestyle accommodation (decreased activity, a cane, high chairs and toilet seats, etc), non-steroidal anti-inflammatory drugs (NSAIDS), anti-arthritics, steroids, various and sundry prescription and non-prescription oral and topical medications and exercise. Randomized controlled trials (RCTS) support exercise for KOA treatment, proven superior to placebo. At least 50% (and periodically up to 90 percent) of KOA patients regularly use NSAIDs. Frequent minor but intermittently serious gastrointestinal and cardiovascular adverse reactions to chronic use of NSAIDS occur, and there is evidence that using exercise/rehabilitation with or without manipulative (MAN) therapy may give safer, similar or equivalent relief. Supported by earlier RCTs, MAN therapy with and without soft tissue and exercise therapy for KOA appears superior to placebo and equal or superior to exercise. Although Chiropractic has conducted and published two RCTs of manipulative therapy for KOA, the profession has not yet conducted an RCT with combined full kinetic chain MAN therapy, soft tissue and rehabilitation versus standard care (rehabilitation or exercise therapy) nor studied optimum dose for various patients. 1). in effect only 1 study of such combined care (MAN therapy, soft tissue and rehabilitation or exercise therapy) exists; 2) more studies of MAN therapy combined with rehabilitation are needed to establish: a). equivalent or b). superior treatment efficacy with full kinetic chain therapy and to c). use 'dose time to response' techniques to study the optimum number of treatments for various patients and (to help determine who will respond and will not respond and why) and d)collect data to develop future cost effective research.

Significant morbidity and occasional mortality from NSAID and drug-related complications and surgery; difficulty in obtaining compliance with prolonged exercise protocols; apparent similar, equivalent or superior outcomes (manipulative therapy with and without, but possibly superior with, combined rehabilitation) in pain relief, mobility and function; the possibility of decreasing falls with their appalling sequela in morbidity, mortality and expense; justifies further research into multimodal manipulative therapy for treatment of KOA. Data suggests such full kinetic chain MAN therapy with rehabilitation may give earlier, effective, less costly outcomes and reflects a common clinical chiropractic approach to KOA. In addition to the knee joint, KOA disability has been demonstrated to be significantly worsened by hip joint dysfunction, for example restricted hip flexion increases KOA pain and dysfunction; and there are similar associations throughout the full kinetic chain for example lumbosacral spine joint dysfunction may increase knee pain and dysfunction. Manipulative therapy applied appropriately to the full, kinetic chain (to the full axial and appendicular skeleton -the spine and extremities) combined with rehabilitation may be a superior treatment for knee OA.

ELIGIBILITY:
Inclusion Criteria:

1. Knee pain and crepitus with active motion and morning stiffness ≤ 30 min ages ≥ 38 and ≤ 80
2. Knee pain and crepitus with active motion and morning stiffness >30 minutes and boney enlargement ages ≥ 38 and ≤ 80
3. Knee pain and no crepitus and boney enlargement ages ≥ 38 and ≤ 80 Note: knee x-rays taken in each case to determine grades (0-4) Kellgren Lawrence x-ray scale - but not required for diagnosis - (and if needed lumbosacral/pelvic, hip, ankle or foot x-rays obtained) see exclusions below)
4. Knee pain (mild to moderate) of 1 year duration and age ≥ 38 and ≤ 80 years of age and able to stand and walk (see informed consent)
5. Diagnosis of concurrent subluxation/joint dysfunction (S/JD) complex a) Diagnosis of S/JD will be supported throughout using the PART(S) system 6).A patient must have a score of ≥720 mm on the WOMAC to be included (≥30%) 7).Additionally, KOA patients, who are + for the Berg Balance Scale (BBS) will be monitored as a subgroup (with OLST and BBS) at all clinic assessments.

Exclusion Criteria:

Rule out: General and internal medical disorders such as significant visual disorders, severe vestibular disorders (i.e., Meniere's), neurological (including Alzheimer's and other degenerative brain and mental disorders, disease and dysfunction) peripheral sensory disorders (severe insulin dependent diabetes), knee and hip joint replacement on side of knee that is treated (case by case otherwise), RA, instability, fracture/ and severe osteoporosis, frank avascular necrosis with or without moderate or severe deformity, lumbar herniated disc and injury, severe balance and proprioception problems (i.e., inability to stand with and/or without marked spinal, knee or hip deformity) etc. Symptoms (moderate to severe) in both knees or hips (case by case), etc. Recent history of meniscal or other knee surgery (not less than 6 months). Severe/constant self reported knee crepitus. Severe loss of knee or hip ROM and or severe deformity (in valgus, varus etc) particularly with instability. Severe depression per Beck Depression Index. Marked or severe fear of chiropractic adjustments/manipulative and or exercise procedures. Breaks for treatment longer than 3-4 weeks depending on each circumstance or merit may be construed as non-compliance and may be excluded.

-

Ages: 38 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2010-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
McMaster Overall Therapy Effectiveness Tool | 15 months
Western Ontario and McMaster Universities Osteoarthritis index | 15 months

SECONDARY OUTCOMES:
Range of Motion | 15 months
  Range of motion of the knee
One Leg Standing Test | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: James W Brantingham, DC, PhD, Principal Investigator — Cleveland Chiropractic College
Locations (2):
- Cleveland Chiropractic College Health Center, Los Angeles, California, United States
- Durban University of Technology, Durban, South Africa

REFERENCES:
- [Result] Deyle GD, Allison SC, Matekel RL, Ryder MG, Stang JM, Gohdes DD, Hutton JP, Henderson NE, Garber MB. Physical therapy treatment effectiveness for osteoarthritis of the knee: a randomized comparison of supervised clinical exercise and manual therapy procedures versus a home exercise program. Phys Ther. 2005 Dec;85(12):1301-17. PMID 16305269
- [Result] Pollard H, Ward G, Hoskins W, Hardy K. The effect of a manual therapy knee protocol on osteoarthritic knee pain: a randomised controlled trial. J Can Chiropr Assoc. 2008 Dec;52(4):229-42. PMID 19066697
- [Result] Hoeksma HL, Dekker J, Ronday HK, Heering A, van der Lubbe N, Vel C, Breedveld FC, van den Ende CH. Comparison of manual therapy and exercise therapy in osteoarthritis of the hip: a randomized clinical trial. Arthritis Rheum. 2004 Oct 15;51(5):722-9. doi: 10.1002/art.20685. PMID 15478147
- [Result] Fish D, Kretzmann H, Brantingham JW, Globe G, Korporaal C, Moen J. A Randomized Clinical Trial to Determine the Effect of Combining a Topical Capsaicin Cream and Knee-Joint Mobilization in the Treatment of Osteoarthritis of the Knee. Journal of the American Chiropractic Association 8-23, August 2008.